CLINICAL TRIAL: NCT02178163
Title: A Study to Assess the Ability to Initiate Therapy in Advanced Non-small Cell Lung Cancer (NSCLC) Patients Based on Genomic Analyses of Tumor Specimens.
Brief Title: Comprehensive Genomic Analysis in Tissue Samples From Patients With Recurrent or Stage IV Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gerold Bepler, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-002; NCI-2014-00913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); W81XWH-11-1-0500 (Other: Dept of Defense); 2014-002 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This study will assess the percentage of advanced NSCLC patients whose tumor samples can undergo genomic analysis and in whom therapy can begin based on the results of this analysis.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ancillary-Correlative (comprehensive genomic analysis) (Experimental): Patients undergo collection of tissue samples for genomic analysis via mass spectrometry, PCR, and microarray. Based on the results of the genomic analysis, patients may begin therapy.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies comprehensive genomic analysis in tissue samples from patients with non-small cell lung cancer that has come back or is stage IV. Comprehensive genomic analysis may identify specific gene mutations (changes in deoxyribonucleic acid [DNA]) and help doctors to tailor treatment to target the specific mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the percentage of advanced non-small cell lung cancer patients in whom therapy can be initiated based on genomic analysis of tumor specimens.

SECONDARY OBJECTIVES:

I. To estimate the percentage of patients in whom genomic analysis can be performed.

II. To assess the progression free survival and response rate in patients who start therapy based on the genomic analyses results.

OUTLINE:

Patients undergo collection of tissue samples for genomic analysis via mass spectrometry, polymerase chain reaction (PCR), and microarray. Based on the results of the genomic analysis, patients may begin therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or recurrent Non-Small Cell Lung Cancer patients who either have archival tissue for genomic analysis or are willing to undergo a new biopsy to obtain tumor tissue for genomic analysis. Patients whose tumor has already undergone genomic analysis will be eligible.
* Zubrod performance status 0-2
* Life expectancy >= 3 months
* Absolute neutrophil count of > 1.5 x 10^9/L
* Platelet count > 100,000 x 10^9/L
* Serum creatinine =< 1.5 times the institutional upper limit of normal (ULN) or calculated creatinine clearance (Cockcroft-Gault formula) of > 45 mL/min
* Serum bilirubin =< 1.5 X ULN
* Transaminases (serum glutamic oxaloacetic transaminase [SGOT] and/or serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times institutional ULN and alkaline phosphatase =< 2.5 times ULN, unless patient has liver metastases and the managing physician believes that the elevation in liver enzymes is only related to the liver metastases
* Laboratory tests should be done within 30 days of enrollment on the trial
* A biopsy of the patient's tumor for genomic profiling is required; this biopsy specimen can be an already obtained diagnostic specimen provided the patient has not received systemic therapy since the biopsy has been obtained and was obtained within 60 days of trial enrollment. The biopsy material cannot be from a tumor site that has been radiated.
* Signed informed consent that details the investigational nature of the study according to institutional and federal guidelines

Exclusion Criteria:

* Patients with concurrent malignancy; patients with prior or concurrent malignancy will be allowed as long as the treating physician considers it unlikely to impact the clinical outcome of the patient
* Serious medical illness including but not limited to uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction or cerebrovascular event with 6 months of registration, history of chronic active hepatitis or history of human immunodeficiency virus (HIV) or an active bacterial infection will not be eligible
* Pregnant or lactating women; female patients of child bearing potential will be informed that if they do enroll on a therapeutic trial, based on the genomic analyses, that they may not be able to enroll on a clinical trial if they are pregnant; all sexually active patients will be informed that patients enrolling on a therapeutic trial have to use contraceptive methods to prevent pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving therapy based on genomic analyses among all eligible patients | Up to 21 days
  Will be estimated with 95% confidence interval (CI) using the Wilson's method.

SECONDARY OUTCOMES:
Overall response rate assessed according to Response Evaluation Criteria in Solid Tumors 1.1 | Up to 2 years
  Response rate will be estimated with 95% Wilson's CI.
Progression free survival (PFS) | Time from the date of start of therapy based on genomic analysis until the date that progressive disease or death whichever is first reported, assessed up to 2 years
  PFS will be estimated and may also be summarized within subgroups using descriptive statistics (Kaplan and Meier) if there are sufficient data.
Overall survival (OS) | From date of registration to up to 2 years
  Not all patients enrolled on the study will receive therapy based on genomic analyses therefore survival will be analyzed for patients who receive therapy based on genomic analyses, for patients who don't receive therapy based on genomic analyses and for the entire patient population. OS will be estimated and may also be summarized within subgroups using descriptive statistics (Kaplan and Meier) if there are sufficient data.

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (11):
- United States (11):
  - KCI at McLaren Bay Region, Bay City, Michigan
  - KCI at Mclaren Bloomfield Hills, Bloomfield Hills, Michigan
  - KCI At McLaren Clarkston, Clarkston, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - KCI at McLaren Flint, Flint, Michigan
  - KCI at McLaren Greater Lansing, Mid Michigan Physicians, Lansing, Michigan
  - KCI at McLaren Lapeer Region, Lapeer, Michigan
  - KCI at McLaren Macomb, Mount Clemens, Michigan
  - KCI at McLaren Central Michigan, Mount Pleasant, Michigan
  - KCI at Northern Michigan, Petoskey, Michigan
  - KCI at McLaren Port Huron, Port Huron, Michigan

IPD SHARING:
Plan to Share IPD: No